CLINICAL TRIAL: NCT03572725
Title: Air Tamponade and Non-supine Positioning in Macular Hole Surgery. A Randomized Controlled Trial.
Brief Title: Air Tamponade and Non-supine Positioning in Macular Hole Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other); Trondheim University Hospital (Other); University Hospital of North Norway (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/785
Record Dates: First submitted 2018-06-11; First posted 2018-06-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-10

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gas tamponade (Active Comparator): Gas as intraocular tamponade.
  Interventions: Procedure: Gas tamponade
- Air tamponade (Experimental): Air as intraocular tamponade.
  Interventions: Procedure: Air tamponade

INTERVENTIONS:
Procedure: Gas tamponade — Removal of intraocular fluid and replacement with intraocular tamponade. No restriction of postoperative positioning with exception to the supine position. A tennis ball is attached to the back of patients at night. This measure will assists them in avoiding the nocturnal supine position.
  Arms: Gas tamponade
Procedure: Air tamponade — Removal of intraocular fluid and replacement with intraocular tamponade. No restriction of postoperative positioning with exception to the supine position. A tennis ball is attached to the back of patients at night. This measure will assists them in avoiding the nocturnal supine position.
  Arms: Air tamponade

SUMMARY:
This is a prospective, multicenter, randomized non-inferiority trial, where the macular hole closure rate with intraocular air tamponade is compared to the closure rate with gas tamponade.The patients are randomized to receive either air or gas (26% SF6) as intraocular tamponade, just prior to the intraocular flushing of the tamponade during the vitrectomy procedure. Postoperatively, the patients adhere to the nonsupine regimen for three days, and the tennis ball technique is used during sleep to enhance patients' positioning compliance.

ELIGIBILITY:
Inclusion Criteria:

* Primary macular hole ≤ 400 μm
* Duration no more than 24 months
* Able to sign informed content
* Signed informed content

Exclusion Criteria:

* Earlier vitreoretinal surgery in present eye
* Secondary macular holes caused by other conditions than vitreomacular traction
* Myopic macular hole, i.e. excessive myopia (more than -6 dioptres)
* Posttraumatic macular hole
* Macular holes secondary to retinal detachment or other retinal diseases
* Surgery under general anesthesia
* Visual acuity below 20/40 in fellow-eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Macular hole closure verified on OCT | 2 - 8 weeks postoperatively
  Macular hole closure verified on OCT after one macular hole intervention

SECONDARY OUTCOMES:
Closure of macular holes ≤ 250 µm | 2 - 8 weeks postoperatively
  Macular hole closure verified on OCT after one macular hole intervention
Closure of macular holes >250 µm and ≤ 400 µm | 2 - 8 weeks postoperatively
  Macular hole closure verified on OCT after one macular hole intervention
Intraocular pressure | First postoperative day
  Standard procedure for assessment of intraocular pressure
Visual acuity | 2 - 8 weeks postoperatively
  Standard procedure for assessment of visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, PhD, Principal Investigator — Helse Stavanger HF
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Department of Ophthalmology, Stavanger
  - University Hospital of North Norway, Tromsø
  - Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindtjorn B, Krohn J, Haugstad M, Stene-Johansen I, Austeng D, Basit S, Fossen K, Varhaug P, Kvaloy JT, Forsaa VA. Air versus Sulfur Hexafluoride Gas Tamponade for Small and Medium-Sized Macular Holes: A Randomized Noninferiority Trial. Ophthalmol Retina. 2022 Sep;6(9):828-834. doi: 10.1016/j.oret.2022.04.003. Epub 2022 Apr 7. PMID 35398546